CLINICAL TRIAL: NCT03437837
Title: Validation of CPS+EG, Neo-Bioscore and Modified Neo-Bioscore Staging System After Preoperative Systemic Therapy of Breast Cancer in Multi-center in China
Brief Title: Validation of the CPS+EG, Neo-Bioscore and Modified Neo-Bioscore Staging Systems After PST of BC in China
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, XU Ling, Associate Chief Physician of Breast Disease Center, Associate Professor, M.D., Peking University First Hospital
Other Study IDs: CPS+EG-NeoBioscore-Modified
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Neoplasm Staging; Estrogen Receptor; Histological Grade; HER2; Prognosis; Predictive Value of Tests
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prognostic assessment after preoperative systemic therapy (PST) plays a vital role in breast cancer patients. The clinical-pathologic staging system incorporating estrogen receptor (ER)-negative disease and nuclear grade 3 tumor pathology (CPS+EG staging system) can effectively predict prognosis after PST. The Neo-Bioscore has been developed by the incorporation of the human epidermal growth factor receptor 2 (HER2) status into the CPS+EG staging system. But in a real world in China, the both staging systems had limits because of trastuzumab administration varied a lot in China from the United States. This retrospective study will validate CPS+EG and Neo-Bioscore system and explored a modified Neo-Bioscore system in multiple centers.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study if he or she meets all of the following criteria:

1. Has operable, histologically confirmed, Stage I, IIA, IIB, IIIA, IIIB or IIIC invasive carcinoma of the breast.
2. Has had neoadjuvant chemotherapy before operation for this breast cancer.
3. Age >=18 to <=75 years old.
4. Has known ER and PR status.
5. Has known HER-2 status.
6. Has known menopausal status.
7. Before PST, Lymph nodes were evaluated by fine needle biopsy (FNB) if the clinically positive, or by sentinel lymph nodes biopsy (SLNB) if the clinically or FNB negative.
8. Has complete surgical resection of the primary breast tumor after PST: either lumpectomy or mastectomy with sentinel lymph node biopsy or axillary dissection, with clear margins for both invasive and ductal carcinoma in situ (DCIS).
9. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
10. Has laboratory values of

    * White blood cell count >3000/mm3
    * Absolute neutrophil count (ANC) ≥1500/mm3
    * Hemoglobin ≥9.0 g/dL
    * Total bilirubin <ULN
    * Serum creatinine ≤1.5 mg/dL
    * Platelet count ≥100,000/mm3
    * ULN = upper limit of normal
11. Has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) and alkaline phosphatase (ALP) within any of the ranges shown below:

    * ALP ≤ upper limits of normal(ULN),and AST or ALT ≤ 5 ULN
    * ULN < ALP ≤2.5 ULN, and AST or ALT ≤ 1.5 ULN
    * 2.5 ULN < ALP ≤5 ULN, and AST or ALT ≤ ULN
12. Has normal cardiac function as evidenced by an left ventricular ejection fraction (LVEF) >50% by echocardiogram (ECHO), Ejection fraction as determined by ECHO must be within normal limits (WNL) by institutional standard.
13. Has no evidence of metastatic disease outside of breast by physical examination and chest x-ray or computed tomography (CT) scan. Other scans if done as needed by the patient [e.g., bone scan; abdominal, chest CT; Positron Emission Tomography (PET) or Positron Emission Tomography-Computed Tomography (PET-CT); ultrasound; or Magnetic Resonance Imaging (MRI)] should indicate no evidence of metastatic disease.
14. Has had baseline bilateral B-type ultrasound，MRI was recommended, but not essential.
15. If fertile, patient has agreed to use an acceptable method of birth control (barrier contraceptive only) to avoid pregnancy duration the study and for a period of 3 months thereafter

Exclusion Criteria:

A patient will be excluded from this study if she meets any of the following criteria:

1. Has bilateral synchronous breast cancer.
2. Has any evidence of metastatic disease: staging work-up, biopsy or physical examination suspicious for malignant disease.
3. Has a history of severe hypersensitivity reaction to chemotherapy drugs or formulation.
4. Has a history of heart failure, uncontrolled angina, severe uncontrolled arrhythmias, pericardial disease, or electrocardiographic evidence of acute ischemic changes.
5. Has peripheral neuropathy >Grade 1.
6. Has had a major organ allograft or condition requiring chronic immunosuppression (ie, kidney, liver, lung, heart, bone marrow transplant, or autoimmune diseases). Patients who have received corneal transplants or cadaver skin or bone transplants are eligible.
7. Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious viral [including clinically defined acquired immune deficiency syndrome (AIDS)], bacterial or fungal infection; or history of uncontrolled seizures, or diabetes, or central nervous system (CNS) disorders deemed by the Treating Physician to be clinically significant, precluding informed consent.
8. Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be human immunodeficiency virus (HIV) positive.
9. Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin, carcinoma in situ of uterine cervix, DCIS), which could affect the diagnosis or assessment of any of the study drugs.
10. Is deemed unable to comply with requirements of study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonmetastatic primary breast cancer patients who were treated with preoperative systemic therapy and surgery and had complete interesting clinicopathological data will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Disease Specific Survival (DSS) | 5 years
  DSS will be calculated from the time of diagnosis to death resulting from breast cancer. Patients still alive at the time of the analysis will be censored using the date they were last known to be alive.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  DFS, defined as the time from the time of post-PST breast cancer surgery to local recurrence following mastectomy, local recurrence in the ipsilateral breast following lumpectomy (invasive or non-invasive), regional recurrence, distant metastasis, contralateral breast cancer (invasive or non-invasive), second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colorectal carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause prior to recurrence or second primary cancer. Patients who have not had any such event at the time of data analysis will be censored at the last date they were known to be event-free.
Overall Survival (OS) | 5 years
  OS will be measured as the time from the date of diagnosis to the date of death. Patients still alive at the time of the analysis will be censored using the date they were last known to be alive.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The 4th Hospital of Hebei medical university, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning, China, Shenyang, Liaoning
  - Xijing Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Second Affiliated Hospital of Shantou University Medical College, Jinan, Shandong

REFERENCES:
- [Derived] Xu L, Liu Y, Fan Z, Jiang Z, Liu Y, Ling R, Zhang J, Yu Z, Jin F, Wang C, Cui S, Wang S, Mao D, Han B, Wang T, Zhang G, Wang T, Guo B, Yu L, Xu Y, Fu F, Liu Z, Wang S, Luo K, Xiang Q, Zhang Z, Liu Q, Zhou B, Liu Z, Ma C, Tong W, Mao J, Duan X, Cui Y. Assessment of CPS + EG, Neo-Bioscore and Modified Neo-Bioscore in Breast Cancer Patients Treated With Preoperative Systemic Therapy: A Multicenter Cohort Study. Front Oncol. 2021 Mar 16;11:606477. doi: 10.3389/fonc.2021.606477. eCollection 2021. PMID 33796452